CLINICAL TRIAL: NCT04630756
Title: A Modular Phase I/II, Open-label, Multicentre Study to Assess AZD4573 in Novel Combinations With Anti-cancer Agents in Patients With Advanced Haematological Malignancies
Brief Title: AZD4573 in Novel Combinations With Anti-cancer Agents in Patients With Advanced Blood Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8230C00002; 2020-001642-18 (EudraCT Number)
Record Dates: First submitted 2020-09-02; First posted 2020-11-16 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Advanced Haematological Malignancies
Keywords: AZD4573; Anti-cancer Agents; Sequential dose-setting and expansion treatment
MeSH Terms: interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1: Part A and Part B (Experimental): Participants will receive intravenous ascending doses of AZD4573 once weekly with oral acalabrutinib twice daily continuously in Part A. For Part A, cohorts 1, 2, and 3 have different target dose levels respectively.
  In Part B, participants will receive the RP2D of AZD4573 from Part A.
  Interventions: Drug: AZD4573; Drug: Acalabrutinib
- Module 2: Part A and Part B (Experimental): Participants will receive AZD4573 as monotherapy for Period 1 and AZD4573 + acalabrutinib as combination therapy for Period 2.
  Part B of Module 2 will be determined from the data emerging from Part A.
  Interventions: Drug: AZD4573; Drug: Acalabrutinib

INTERVENTIONS:
Drug: AZD4573 — AZD4573 will be administered as an absolute (flat) dose, 2-hour (± 15 minutes) IV infusion once weekly (as monotherapy for Module 2 only) and in combination with orally administered acalabrutinib twice daily continuously. For both Part A and Part B of this study, Cycle 1 consists of 5 weeks, with a dose ramp-up. Subsequent cycles are 21 days (3 weeks) with once weekly dosing of AZD4573 in combination with acalabrutinib twice daily continuously (in Module 1 and Module 2, period 2).
  Other Names: AZ13810325
Drug: Acalabrutinib — Oral Acalabrutinib capsule will be administered twice daily continuously from Day 1 of Cycle 1 Week 1 in combination with AZD4573.
  Other Names: ACP-196 /Calquence

SUMMARY:
This is a modular, multicentre, open-label, non-randomised, Phase I/II, dose-setting and expansion study including an intra-participants dose ramp up. AZD4573 will be administered intravenously, in novel combinations with anti-cancer agents, to participants with relapsed/refractory (r/r) haematological malignancies.

DETAILED DESCRIPTION:
In Module 1 Part A (dose-setting), this study module will enrol participants with r/r Diffuse large B-cell lymphoma (DLBCL) or r/r Marginal zone lymphoma (MZL) who have failed prior therapy(ies), are not eligible for curative treatment options, for whom there is no standard therapy available, and will initially explore once weekly administration of AZD4573 at up to three target dose levels in combination with oral acalabrutinib 100 mg twice daily. The primary objective of Part A will be to identify the maximum tolerated dose and/or Recommended Phase II dose (RP2D) for further evaluation in Part B. A 5-week DLT-assessment period will incorporate the whole of Cycle 1 in Part A, including the dose ramp up and the first 3 weeks at the target dose. In Module 1 Part B (expansion), separate expansion cohorts for participants with Germinal Centre B-cell (GCB) and non-GCB DLBCL subtypes will be opened at the RP2D.

In Module 2, this study module will enroll participants with r/r Mantle Cell Lymphoma (MCL) who have failed at least one line of prior therapy, are not eligible for curative treatment options. Module 2, Part A consist of AZD4573 monotherapy (Period 1) followed by AZD4573 + acalabrutinib combination treatment (Period 2). Period 1: AZD4573 will be administered weekly (12 mg, infusion). Period 2: AZD4573 (RP2D from Module 1) will be administered (weekly) in combination with oral acalabrutinib 100 mg twice daily. Cycle 1 of each dosing period has a duration of 5 weeks; subsequent cycles have a duration of 3 weeks. The AZD4573 monotherapy (Period 1) includes an intra-patient ramp up; participants will receive AZD4573 at Cycle 1 Week 1, Cycle 1 Week 2, and Cycle 1 Week 3 in 3 dose escalation manner (6, 9 and 12 mg respectively). Part A, Period 1 of Module 2 aims to confirm the AZD4573 monotherapy RP2D in MCL participants. In Period 2, the safety and tolerability of the RP2D of AZD4573 + acalabrutinib established in Module 1 will be assessed in participants with MCL. The study design of Part B of Module 2 will be determined from the data emerging from Part A.

ELIGIBILITY:
Inclusion Criteria - Core

* Participant must be ≥ 18 years of age at the time of signing the informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Must have received at least one prior line of therapy for the treatment of current disease and a clinical study is the best option for next treatment based on prior response and/or tolerability.
* Documented active disease requiring treatment that is r/r defined as: Recurrence of disease after response to at least one prior line(s) of therapy or Progressive disease after completion of or on the treatment regimen preceding entry into the study or Disease that did not achieve an objective response (overall response of CR or PR).
* Adequate haematological function.
* Adequate organ function at Screening.
* Uric acid level < upper limit of normal (ULN).

Inclusion Criteria - Module 1

- Participants with histologically confirmed, r/r DLBCL, or r/r MZL, for whom a clinical study is the best option for next treatment based on response and/or tolerability to prior lines of therapy.

PART A

• Participants with r/r DLBCL, including subtypes such as DLBCL not otherwise specified [NOS], high-grade B cell lymphoma [HGBCL], primary mediastinal large B-cell lymphoma [PMBCL], or large B cell lymphoma transformed from indolent B-cell lymphomas (including but not limited to Richter Syndrome, transformed Follicular Lymphoma, transformed MZL), or r/r MZL: participants with r/r MZL are eligible as well. In case fresh tumor biopsy is not available, archival tumor samples are acceptable, if done with 24 months

PART B • Participants with r/r de novo r/r DLBCL only, fresh tumor biopsy, done at screening or within 60 days before planned 1st dosing, unless there was any anticancer treatment given after tumor biopsy, but prior initiated study treatment.

* Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy.
* Participants must have failed at least two prior therapies for the treatment of current disease. Participants shall not be eligible for curative treatment options, and have no standard therapy available (including CAR-T cell therapy).
* Adequate haematologic function at screening: No growth factor support within 14 days prior to the date of the screening laboratory assessment; No transfusions within 7 days prior to the date of the screening laboratory assessment.
* Optional tumour biopsy on study: Participants are also encouraged to consent to and undergo an optional tumour biopsy at disease progression to support correlative biomarker studies.
* All participants must be willing and able to provide mandatory baseline bone marrow biopsy/aspirate.

Inclusion Criteria - Module 2

- Participants with histologically confirmed r/r MCL for whom a clinical study is the best option (in the opinion of the investigator) for next treatment based on response and/or tolerability to prior lines of therapy.

PART A

* Participants with r/r MCL:

  * Diagnosis must be confirmed by biopsy and be immunohistologically characterised.
  * Tumour tissue must also be available for sending to AstraZeneca for pathology testing.
* Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy
* Participants must have failed at least one prior therapy for the treatment of current disease and not be eligible for treatment with curative intent (e.g. allogenichaematopoietic cell transplantation [HCT]). Eligible participants include both BTKi-naïve and BTKi-exposed.
* Adequate haematologic function at screening: No growth factor support within 14 days prior to the date of the screening laboratory assessment; No transfusions within 7 days prior to the date of the screening laboratory assessment.
* Optional tumour biopsy on study: Participants are also encouraged to consent to and undergo an optional tumour biopsy at disease progression to support correlative biomarker studies.
* All participants must be willing and able to provide mandatory baseline bone marrow biopsy/aspirate.

Exclusion Criteria - Core

* Participants with non-secretory myeloma.
* With the exception of alopecia, any unresolved non-haematological toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment.
* Presence of, or history of, central nervous system (CNS) lymphoma, leptomeningeal disease, or spinal cord compression.
* History of prior non-haematological malignancy except for the following: Malignancy treated with curative intent and with no evidence of active disease for >1 year before Screening and felt to be at low risk for recurrence by treating physician; Adequately treated lentigo maligna melanoma without evidence of disease or adequately controlled non-melanomatous skin cancer; Adequately treated carcinoma in situ without current evidence of disease.
* Any evidence of severe or uncontrolled systemic disease (eg, severe hepatic impairment, interstitial lung disease), or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension, history of, or active, bleeding diatheses or uncontrolled active systemic fungal, bacterial, viral, or other infection, or IV anti infective treatment within two weeks before first dose of study drug.
* Known history of infection with human immunodeficiency virus (HIV).
* Serologic status reflecting active hepatitis B or C infection.
* Any of the following cardiac criteria: Resting QT interval corrected using Fridericia's formula (QTcF) ≥ 470 msec obtained from a single electrocardiogram (ECG); any clinically important abnormalities in rhythm (except for participants with a pacemaker in place), conduction or morphology of resting ECG); any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age. Concomitant medications known to prolong QTc should be used with caution and cannot be used starting with the first dose of study drug and through the DLT-assessment period (Part A) or during the scheduled ECG assessments.
* History of severe allergic or anaphylactic reactions to BH3 mimetics or history of hypersensitivity to active or inactive excipients of study treatment.
* Documented confirmation and ongoing treatment of adrenal gland insufficiency or pancreatitis.
* History, within the previous 6 months prior to first dose, of: coronary artery bypass graft; angioplasty; vascular stent; myocardial infarction; angina pectoris; congestive heart failure (New York Heart Association Class ≥ 2); ventricular arrhythmias requiring continuous therapy; atrial fibrillation, which is judged as uncontrolled by the treating physician; haemorrhagic or thrombotic stroke, including transient ischaemic attacks or any other CNS bleeding.

Exclusion Criteria: Module 1

* Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal function, stomach resection, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, bowel obstruction, or gastric restrictions and bariatric surgery.
* Prior use of standard anti-lymphoma therapy or radiation therapy within 14 days of receiving the first dose of study treatment.
* Requires treatment with strong CYP3A inhibitors or inducers.
* Requires treatment with proton-pump inhibitors. Participants receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrolment to this study.
* Serologic status reflecting active hepatitis B or C infection.
* Active Cytomegalovirus (CMV) infection.
* Requires or receiving therapeutic anticoagulants, with the exception of short-acting heparins, within 7 days of first dose of study treatment. Novel oral anticoagulants are allowed except for the initial high dose treatment period.
* Participants on dual antiplatelet and therapeutic anticoagulant therapy.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists.
* History of or ongoing confirmed progressive multifocal leukoencephalopathy

Exclusion Criteria: Module 2

* Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal function, stomach resection, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery.
* Prior use of standard anti-lymphoma therapy or radiation therapy within 14 days of receiving the first dose of study treatment.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists.
* Requires treatment with strong CYP3A inhibitors or inducers.
* Requires treatment with proton-pump inhibitors. Participants receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrolment to this study.
* Serologic status reflecting active hepatitis B or C infection.
* Active CMV infection.
* Requires or receiving therapeutic anticoagulants, with the exception of short-acting heparins, within 7 days of first dose of study treatment. Novel oral anticoagulants are allowed except for the initial high dose treatment period.
* Participants on dual antiplatelet and therapeutic anticoagulant therapy.
* History of or ongoing confirmed progressive multifocal leukoencephalopathy

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (4):
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
- Australia (2):
  - Research Site, Clayton
  - Research Site, Nedlands
- Research Site, Québec, Quebec, Canada
- Research Site, Lille, France
- Ireland (2):
  - Research Site, Dublin
  - Research Site, Galway
- Research Site, Krakow, Poland
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Palma de Mallorca
- Research Site, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D8230C00002_CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8230C00002&attachmentIdentifier=d1eaa448-66c8-4499-9d93-37f6456d6631&fileName=D8230C00002_CSP_redacted.pdf&versionIdentifier=
- See also: D8230C00002_CSR Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8230C00002&attachmentIdentifier=1b416912-406c-49e4-aa2c-5e1bff487544&fileName=D8230C00002_CSR_Synopsis_redacted.pdf&versionIdentifier=
- See also: D8230C00002_Statistical Analysis Plan_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8230C00002&attachmentIdentifier=6c69478f-31ac-4bdb-a9ca-dda138ca2ad6&fileName=D8230C00002_Statistical_Analysis_Plan_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 17 February 2021 to 08 September 2023. Module 1 was conducted at 17 study centers in 10 countries. Module 2 was conducted at 2 sites in the United States.
Pre-assignment Details: The screening period was of 30 days for both parts of the study. Informed Consent Form (ICF) was signed prior to screening procedures. All the study assessments were performed as per the schedule of assessment. Participants who met the eligibility criteria were randomized to study intervention in addition to receiving background local standard of care therapy.
Groups:
- Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID: Participants received AZD4573 9 mg as Intravenous (IV) infusion once weekly with acalabrutinib 100 mg twice daily.
- Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID: Participants received AZD4573 dose expansion to RP2D 12 mg as IV infusion once weekly with acalabrutinib 100 mg twice daily.
- Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID: Participants received AZD4573 12 mg monotherapy until progression and thereafter received a combination regimen of AZD4573 12 mg once weekly and acalabrutinib 100 mg twice daily.
Period: Module 1 Part A: AZD4573 9 mg
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID
Started | 9 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Ongoing subjects in Post Trial Access Program | 1 | 0 | 0
Period: Module 1 Part B: AZD4573 12 mg
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID
Started | 0 | 28 | 0
Completed | 0 | 28 | 0
Not Completed | 0 | 0 | 0
Period: Module 2 Period 1: AZD4573 Monotherapy
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID
Started | 0 | 0 | 3
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0
Period: Module 2 Period 2: AZD4573 Combination
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID
Started | 0 | 0 | 3
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received any amount of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID | Total
Number analyzed (Participants) | 9 | 28 | 3 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 17 | 3 | 27
  >=65 years | 2 | 11 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 0 | 14
  Male | 5 | 18 | 3 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 8 | 0 | 10
  White | 6 | 17 | 2 | 25
  Not Reported | 1 | 1 | 0 | 2
  Missing | 0 | 2 | 0 | 2
  Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Module 1: Number of Participants With Adverse Events
Description: Safety and tolerability of AZD4573 in combination with acalabrutinib was assessed.
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Population: The safety analysis set included all participants who received any amount of AZD4573 and/or acalabrutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 9 | 28
Participants
  Any adverse event (AE) | 9 | 28
  Any serious adverse event (SAE) | 4 | 16

2. Primary Outcome: Module 2: Number of Participants With Adverse Events
Description: Assessed safety and confirmed the RP2D of AZD4573 monotherapy in MCL participants and assessed the safety and tolerability of AZD4573 in combination with acalabrutinib in participants administered AZD4573 monotherapy.
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Population: The safety analysis set included all participants who received any amount of AZD4573 and/or acalabrutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID
Number analyzed (Participants) | 3
Participants
  Any AE | 3
  Any SAE | 1

3. Secondary Outcome: Module 1: Complete Response (CR) Rate
Description: CR is defined as no detectable evidence of tumor, according to the revised response criteria for malignant lymphoma.
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Population: The response evaluable analysis set included participants dosed with AZD4573 or acalabrutinib with a baseline tumour assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants with response
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 9 | 28
Percentage of participants with response | 11.1 [0.3 to 48.2] | 21.4 [8.3 to 41.0]

4. Secondary Outcome: Module 1: Duration of Response (DoR)
Description: DoR, defined as the time from the first objective response of CR or PR to the time of documented disease progression or death due to any cause, whichever occurs first.
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 9 | 28
Months | 4.4 [4.1 to NA] — Values are not calculated due to insufficient number of participants with events. | 3.3 [1.2 to 6.2]

5. Secondary Outcome: Module 1: Progression Free Survival (PFS)
Description: PFS, defined as the time from first dose date to documented disease progression, or death from any cause, whichever occurs first
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Population: The full analysis set included all participants who received any amount of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 9 | 28
Months | 2.1 [0.30 to 6.44] | 2.8 [1.91 to 3.98]

6. Secondary Outcome: Module 1: Overall Survival (OS)
Description: OS, defined as the time from first dose until the date of death from any cause.
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Population: The full analysis set included all participants who received any amount of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 9 | 28
Months | NA [3.52 to NA] — Values are not calculated due to insufficient number of participants with events. | 8.8 [3.91 to NA] — Values are not calculated due to insufficient number of participants with events.

7. Primary Outcome: Module 1: Overall Response Rate (ORR) of AZD4573 in Combination With Acalabrutinib
Description: Overall response rate (ORR), defined as the proportion of participants who have a tumour response (complete response [CR] and partial response [PR]).
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants with response
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 9 | 28
Percentage of participants with response | 44.4 [13.7 to 78.8] | 50.0 [30.6 to 69.4]

8. Secondary Outcome: Module 1: Cmax of AZD4573
Description: Maximum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered (Cmax).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: The pharmacokinetic analysis set included all dosed patients with reportable plasma concentrations and no important adverse events or protocol deviations that may impact PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 9 | 12
nanograms per milliliter (ng/mL)
  Cycle 1 Week 1 Day 1 | 164.2 (469.0) | 112.6 (70.20)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 2 Day 1 | 235.7 (359.3) | 185.3 (50.61)
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 8 | 11
  Cycle 1 Week 3 Day 1 | 337.8 (194.3) | 270.8 (38.61)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 6 | 9
  Cycle 2 Week 1 Day 1 | 643.1 (578.0) | 294.6 (48.83)

9. Secondary Outcome: Module 1: Cmax of Acalabrutinib
Description: as for outcome 8
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 7 | 11
nanograms per milliliter (ng/mL)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 1 Day 1 | 219.9 (66.94) | 306.1 (76.06)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 10
  Cycle 1 Week 2 Day 1 | 209.8 (45.79) | 322.7 (95.53)
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 7 | 10
  Cycle 1 Week 3 Day 1 | 232.1 (74.77) | 274.2 (78.98)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 5 | 8
  Cycle 2 Week 1 Day 1 | 217.5 (100.8) | 256.7 (67.75)

10. Secondary Outcome: Module 1: Cmax of ACP-5862
Description: as for outcome 8
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 7 | 11
nanograms per milliliter (ng/mL)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 1 Day 1 | 199.2 (129.3) | 250.2 (78.12)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 10
  Cycle 1 Week 2 Day 1 | 382.1 (51.58) | 288.0 (63.26)
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 7 | 10
  Cycle 1 Week 3 Day 1 | 320.8 (35.92) | 282.9 (55.76)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 5 | 8
  Cycle 2 Week 1 Day 1 | 304.6 (79.28) | 251.8 (45.54)

11. Secondary Outcome: Module 1: AUClast of AZD4573
Description: Area under the plasma concentration time curve from zero to the time of the last measurable concentration (AUClast).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 8 | 12
hours*nanogram per milliliter (h*ng/mL)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 12
  Cycle 1 Week 1 Day 1 | 532.9 (164.5) | 561.3 (60.83)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 2 Day 1 | 845.3 (134.8) | 929.0 (55.85)
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 8 | 11
  Cycle 1 Week 3 Day 1 | 1273 (127.7) | 1697 (62.55)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 6 | 9
  Cycle 2 Week 1 Day 1 | 1939 (330.9) | 1439 (90.63)

12. Secondary Outcome: Module 1: AUClast of Acalabrutinib
Description: Area under the plasma concentration time curve from zero to the time of the last measurable concentration (AUClast).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 7 | 11
hours*nanogram per milliliter (h*ng/mL)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 1 Day 1 | 493.9 (58.91) | 631.4 (69.98)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 10
  Cycle 1 Week 2 Day 1 | 520.9 (46.04) | 638.2 (81.66)
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 7 | 10
  Cycle 1 Week 3 Day 1 | 475.9 (45.57) | 570.7 (67.75)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 5 | 8
  Cycle 2 Week 1 Day 1 | 481.8 (58.39) | 424.5 (162.8)

13. Secondary Outcome: Module 1: AUClast of ACP-5862
Description: Area under the plasma concentration time curve from zero to the time of the last measurable concentration (AUClast).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 7 | 11
hours*nanogram per milliliter (h*ng/mL)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 1 Day 1 | 673.9 (93.89) | 870.8 (68.73)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 10
  Cycle 1 Week 2 Day 1 | 1173 (48.03) | 1135 (54.95)
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 7 | 10
  Cycle 1 Week 3 Day 1 | 1204 (36.24) | 1093 (54.50)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 5 | 8
  Cycle 2 Week 1 Day 1 | 941.9 (102.5) | 849.3 (60.56)

14. Secondary Outcome: Module 1: AUCinf of AZD4573
Description: Area under the plasma concentration time curve from zero extrapolated to infinity (AUCinf).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 5 | 9
h*ng/mL
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 1 | 4
  Cycle 1 Week 1 Day 1 | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) is not calculable for a single participant. | 640.5 (15.33)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 4 | 6
  Cycle 1 Week 2 Day 1 | 1188 (160.1) | 847.4 (68.22)
  Cycle 1 Week 3 Day 1 | 1588 (169.6) | 1736 (67.09)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 4 | 5
  Cycle 2 Week 1 Day 1 | 4672 (162.9) | 1853 (29.55)

15. Secondary Outcome: Module 1: AUCinf of Acalabrutinib
Description: Area under the plasma concentration time curve from zero extrapolated to infinity (AUCinf).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 3 | 5
h*ng/mL
  Cycle 1 Week 1 Day 1 | 600.1 (34.99) | 501.3 (58.03)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Module 1: AUCinf of ACP-5862
Description: Area under the plasma concentration time curve from zero extrapolated to infinity (AUCinf).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 2 | 4
h*ng/mL
  Cycle 1 Week 1 Day 1 | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) values is not calculated for less than three participants. | 935.2 (38.81)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Module 1: Tmax of AZD4573
Description: Time to reach peak or maximum observed concentration following drug administration (tmax).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 8 | 12
Hours (h)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 12
  Cycle 1 Week 1 Day 1 | 1.992 [0.750 to 4.17] | 2.083 [1.00 to 10.5]
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 2 Day 1 | 1.892 [1.00 to 3.00] | 2.033 [1.05 to 2.15]
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 8 | 11
  Cycle 1 Week 3 Day 1 | 2.192 [0.933 to 3.32] | 2.000 [1.03 to 2.15]
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 6 | 9
  Cycle 2 Week 1 Day 1 | 2.067 [1.00 to 2.22] | 2.083 [1.85 to 3.63]

18. Secondary Outcome: Module 1: Tmax of Acalabrutinib
Description: Time to reach peak or maximum observed concentration following drug administration (tmax).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 7 | 11
Hours (h)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 1 Day 1 | 1.242 [1.02 to 3.80] | 1.117 [0.933 to 2.65]
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 9
  Cycle 1 Week 2 Day 1 | 2.017 [1.00 to 4.52] | 1.133 [0.950 to 11.6]
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 7 | 10
  Cycle 1 Week 3 Day 1 | 1.233 [1.00 to 3.17] | 1.433 [0.850 to 4.00]
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 5 | 7
  Cycle 2 Week 1 Day 1 | 1.933 [1.03 to 5.75] | 1.200 [0.833 to 2.25]

19. Secondary Outcome: Module 1: Tmax of ACP-5862
Description: Time to reach peak or maximum observed concentration following drug administration (tmax).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 7 | 11
Hours (h)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 6 | 11
  Cycle 1 Week 1 Day 1 | 3.067 [1.02 to 7.00] | 1.117 [0.933 to 7.08]
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 6 | 9
  Cycle 1 Week 2 Day 1 | 2.075 [1.08 to 7.52] | 2.117 [1.05 to 11.6]
  Cycle 1 Week 3 Day 1: number analyzed (Participants) | 7 | 10
  Cycle 1 Week 3 Day 1 | 1.233 [1.00 to 4.58] | 1.892 [0.850 to 4.00]
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 5 | 7
  Cycle 2 Week 1 Day 1 | 2.167 [2.05 to 8.92] | 2.117 [0.917 to 4.13]

20. Secondary Outcome: Module 1: t1/2 of AZD4573
Description: Time taken for half the initial dose of drug administered to be eliminated from the body (t1/2).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 5 | 10
Hours (h)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 1 | 5
  Cycle 1 Week 1 Day 1 | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) is not calculable for a single participant. | 3.692 (37.98)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 4 | 7
  Cycle 1 Week 2 Day 1 | 3.364 (43.80) | 5.407 (73.47)
  Cycle 1 Week 3 Day 1 | 4.465 (42.28) | 6.177 (30.16)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 4 | 5
  Cycle 2 Week 1 Day 1 | 6.508 (30.61) | 5.808 (25.52)

21. Secondary Outcome: Module 1: t1/2 of Acalabrutinib
Description: Time taken for half the initial dose of drug administered to be eliminated from the body (t1/2).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 6 | 6
Hours (h)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 3 | 5
  Cycle 1 Week 1 Day 1 | 1.332 (22.01) | 1.108 (12.06)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 3 | 6
  Cycle 1 Week 2 Day 1 | 1.383 (49.15) | 1.274 (25.09)
  Cycle 1 Week 3 Day 1 | 1.238 (20.93) | 1.546 (38.08)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 2 Week 1 Day 1 | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) values was not calculated for less than three participants. | 1.398 (32.20)

22. Secondary Outcome: Module 1: t1/2 of ACP-5862
Description: Time taken for half the initial dose of drug administered to be eliminated from the body (t1/2).
Time Frame: Cycle 1 (5 weeks in total) on Day 1 of Week 1, 2 and 3, and Cycle 2 (3 weeks in total) on Day 1 of Week 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID
Number analyzed (Participants) | 5 | 6
Hours (h)
  Cycle 1 Week 1 Day 1: number analyzed (Participants) | 2 | 5
  Cycle 1 Week 1 Day 1 | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) is not calculated due to insufficient number of participants. | 2.568 (33.27)
  Cycle 1 Week 2 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 1 Week 2 Day 1 | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) values is not calculated for less than three participants. | 3.021 (47.65)
  Cycle 1 Week 3 Day 1 | 2.650 (34.68) | 3.557 (38.06)
  Cycle 2 Week 1 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 2 Week 1 Day 1 |  | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) values is not calculated for less than three participants.

ADVERSE EVENTS:
Time Frame: From Screening (Day -30 to Day -1) until disease progression or survival until death (approximately 2.5 years)
Arm/Group | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID
All-Cause Mortality (participants affected / at risk) | 4/9 | 16/28 | 0/3
Serious Adverse Events (participants affected / at risk) | 4/9 | 16/28 | 2/3
Other Adverse Events (participants affected / at risk) | 9/9 | 28/28 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID (N=9) | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID (N=28) | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID (N=3)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1 Part A: AZD4573 9 mg + 100g Acalabrutinib BID (N=9) | Module 1 Part B: AZD4573 12 mg + 100g Acalabrutinib BID (N=28) | Module 2 Period 1 + 2: AZD4573 12 mg Monotherapy + Combination BID (N=3)
COVID-19 (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lip neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 14 (23) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (86) | 25 (126) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (11) | 16 (46) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 8 (9) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (4) | 1 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 8 (14) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 7 (14) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 6 (13) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 5 (7) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 6 (8) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Scintillating scotoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (6) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (7) | 14 (32) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (7) | 19 (33) | 2 (2)
Saliva altered (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 11 (19) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 3 (9) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Application site erosion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 11 (12) | 2 (2)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 6 (6) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (6) | 15 (46) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (12) | 15 (55) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (5) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 4 (5) | 1 (2)
Fibrin D dimer increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 3 (6) | 0 (0)
Glutamate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 5 (6) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the overall AZD4573 development programme being discontinued as part of a strategic portfolio decision, available data analyzed for this study is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT04630756/Prot_006.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04630756/SAP_007.pdf